CLINICAL TRIAL: NCT02181660
Title: A Phase 1 Open-label, Dose-escalation Study Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP2215 in Japanese Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of ASP2215 in Japanese Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0102
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML; Acute myeloid leukemia; Gilteritinib; ASP2215
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation Cohort (Experimental): ASP2215
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: Gilteritinib — oral
  Other Names: ASP2215

SUMMARY:
The objectives of this study are to determine the safety and tolerability of ASP2215 as well as the maximum tolerated dose (MTD) based on the onset of dose limiting toxicity (DLT) and/or determine the recommended dose (RD) of ASP2215 for the next phase in subjects with relapsed or treatment-refractory acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This study will be conducted to determine the safety, tolerability, PK, PD, and efficacy of single and repeated oral dosing of ASP2215 once daily in patients with relapsed or refractory AML. After the determination of the MTD and/or RD, an expansion cohort might be set to further investigate the safety and efficacy of ASP2215.

This study will consist of a single-dose period (Cycle 0, 2 days) and a repeated-dose period (Cycle 1 and subsequent cycles, each cycle consisting of 28 days). The enrolled subjects will orally receive their assigned single dose in Cycle 0 (Day -2), followed by a 2-day observation period (dosing day inclusive). In Cycle 1 and subsequent cycles (one cycle is defined as 28 days), the subjects will receive oral ASP2215 once daily repeatedly until one of the discontinuation criteria is met. Another dosing regimen may be considered such as dosing twice daily based on the safety and PK data that will become available.

In this study, the Bayesian-Continual Reassessment Method (hereinafter, Bayesian-CRM) will be used as a reference for dose-escalation procedures, and based on the onset of DLTs, the RD level of the subsequent cohort will be set higher or lower. DLTs will be assessed during Cycle 0 and Cycle 1 (30 days).

ASP2215 may be escalated by one dose level if the subject meets the criteria at the end of each cycle after Cycle 1 and the investigator/sub-investigator judges escalation of ASP2215 is of clinical benefit. Dose reduction of ASP2215 will be considered if study drug-related toxicities are observed in a subject.

ELIGIBILITY:
Inclusion Criteria:

* Subject is defined as morphologically documented primary or secondary acute myeloid leukemia (AML) according to the World Health Organization (WHO) criteria (2008) and fulfills one of the following:

  * Refractory to prior induction chemotherapy
  * Relapsed after achieving remission with prior therapy
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Subject's interval from prior treatment to the time of study drug administration is at least 14 days for antineoplastic agents other than ASP2215 (except for hydroxyurea, which is given to control blast cells).
* Subject's interval from prior treatment to the time of study drug (ASP2215) administration is at least 5 half-lives (if the half-life is unknown, 14 days) for other investigational products or drugs used for immunosuppressive therapy posthematopoietic stem cell transplantation (HSCT).

Exclusion Criteria:

* Subject was diagnosed with acute promyelocytic leukemia (APL).
* Subject has breakpoint cluster region-abelson (BCR-ABL)-positive leukemia (chronic myelogenous leukemia in blast crisis)
* Subject has active malignant tumors other than AML or myelodysplastic syndrome (MDS)
* Subject has persistent non-hematological toxicities of ≥ Grade 2 (CTCAE v4), with symptoms and objective findings, due to prior AML treatment (including chemotherapy, kinase inhibitors, immunotherapy, investigational products, radiation therapy, and surgery)
* Subject has received hematopoietic stem cell transplant (HSCT) and falls under either of the following:

  * Is within 2 months of transplant
  * Has persistent and clinically significant graft-versus-host disease requiring treatment
  * Has persistent non-hematological toxicities of ≥ Grade 2 related to the transplant
* Subject has clinically active central nervous system leukemia
* Subject has disseminated intravascular coagulation (DIC)
* Subject has had major surgery within 28 days prior to the first study drug administration
* Subject has had radiation therapy within 28 days prior to the first study drug administration
* Subject has congestive heart failure of NYHA class 3 or 4, or subject with a past history of congestive heart failure of NYHA class 3 or 4 and in whom echocardiogram or Multiple Gate Acquisition (MUGA) scan performed within 3 months prior to screening or at screening showed a left ventricular ejection fraction (LVEF) of < 45%.
* Subject requires treatment with concomitant drugs that are strong inhibitors or inducers of CYP3A4 or of P-gp with such exceptions of antibiotics, antifungals, and antivirals that are considered absolutely essential for prevention or treatment of infections and for which the physician judged that there are no interchangeable drugs.
* Subject requires treatment with concomitant drugs that target serotonin 5HT1R or 5HT2BR receptors or sigma nonspecific receptors, with the exception of drugs that are considered absolutely essential for treatment of the subject.
* Subject has an active uncontrollable infection
* Subject is known to have human immunodeficiency virus (HIV) infection
* Subject has active hepatitis B or C or other active hepatic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-06-27 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability assessed through adverse events to determine maximum tolerated dose | Up to 17 months

SECONDARY OUTCOMES:
Response Rate | Up to 16 months
  Response Rate includes following parameters; CR rate, composite CR [CR + CRp + CRi] rate, overall response rate [CRc + PR], duration of response
Pharmacokinetics of ASP2215 in plasma: AUCinf | Cycle 0 Day -2 through Cycle 1 Day 1
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity
Pharmacokinetics of ASP2215 in plasma: AUClast | Cycle 0 Day -2 through Cycle 1 Day 1
  Area under the concentration-time curve from the time of dosing to the last measurable concentration
Pharmacokinetics of ASP2215 in plasma: AUC24 | Cycle 0 Day -2 through Cycle 1 Day 1
  Area under the plasma concentration time curve from time 0 to 24 hours
Pharmacokinetics of ASP2215 in plasma: AUC48 | Cycle 0 Day -2 through Cycle 1 Day 1
  Area under the plasma concentration time curve from time 0 to 48 hours
Pharmacokinetics of ASP2215 in plasma: Cmax | Cycle 0 Day -2 through Cycle 1 Day 1 and Cycle 1 Day 28
  Maximum concentration
Pharmacokinetics of ASP2215 in plasma: C24 | Cycle 0 Day -2 through Cycle 1 Day 1 and Cycle 1 Day 28
  Concentration at 24 hours
Pharmacokinetics of ASP2215 in plasma: CLF | Cycle 0 Day -2 through Cycle 1 Day 1 and Cycle 1 Day 28
  Oral clearance
Pharmacokinetics of ASP2215 in plasma: Lambda z | Cycle 0 Day -2 through Cycle 1 Day 1
  Terminal first order elimination rate constant
Pharmacokinetics of ASP2215: tmax | Cycle 0 Day -2 through Cycle 1 Day 1 and Cycle 1 Day 28
  Time to attain Cmax
Pharmacokinetics of ASP2215 in plasma: t1/2 | Cycle 0 Day -2 through Cycle 1 Day 1
  Apparent terminal elimination half-life
Pharmacokinetics of ASP2215 in plasma: Vz/F | Cycle 0 Day -2 through Cycle 1 Day 1
  Apparent volume of distribution during the terminal elimination phase after oral dosing
Pharmacokinetics of ASP2215 in plasma: AUCtau | Cycle 1 Day 28
  Area under the plasma concentration time curve during a dosing interval
Pharmacokinetics of ASP2215 in plasma: PTR | Cycle 1 Day 28
  Peak-trough ratio
Pharmacokinetics of ASP2215 in plasma: Rac(AUC) | Cycle 1 Day 28
  Accumulation ratio calculated using the area under the concentration-time curve
Pharmacokinetics of ASP2215 in plasma: Rac(Cmax) | Cycle 1 Day 28
  Accumulation ratio calculated using the maximum concentration
Pharmacokinetics of ASP2215 in plasma: Rac derived t1/2 | Cycle 1 Day 28
  t1/2 derived from accumulation index
Pharmacokinetics of ASP2215 in plasma: Ctrough | Cycle 1 Day 8, Day 15, Day 22, Day 28 and Day 29
  Plasma trough concentration
Pharmacokinetics of ASP2215 in urine: Ae24 | Cycle 0 Day -2 through Cycle 1 Day 1
  Amount of drug excreted in urine from time 0 to 24 hours
Pharmacokinetics of ASP2215 in urine: Ae48 | Cycle 0 Day -2 through Cycle 1 Day 1
  Amount of drug excreted in urine from time 0 to 48 hours
Pharmacokinetics of ASP2215 in urine: Ae24% | Cycle 0 Day -2 through Cycle 1 Day 1
  Fraction of drug excreted into urine from time 0 to 24 hours as % of dose
Pharmacokinetics of ASP2215 in urine: Ae48% | Cycle 0 Day -2 through Cycle 1 Day 1
  Fraction of drug excreted into urine from time 0 to 48 hours as % of dose
Pharmacokinetics of ASP2215 in urine: CLR | Cycle 0 Day -2 through Cycle 1 Day 1 and Cycle 1 Day 28
  Renal clearance
Pharmacokinetics of ASP2215 in urine: Aetau | Cycle 1 Day 28
  Amount of drug excreted in urine during a dosing interval
Pharmacokinetics of ASP2215 in urine: Aetau % | Cycle 1 Day 28
  Fraction of drug excreted in urine during a dosing interval

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Site JP00002, Aichi
  - Site JP00003, Fukuoka
  - Site JP00001, Gunma
  - Site JP00004, Tokyo
  - Site JP00005, Tokyo

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=283